CLINICAL TRIAL: NCT00266877
Title: A Phase 2 Study of HKI-272 In Subjects With Advanced Non-Small Cell Lung Cancer
Brief Title: Study Evaluating the Safety Of HKI-272 (Neratinib) In Subjects With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3144A1-200; B1891037
Record Dates: First submitted 2005-12-16; First posted 2005-12-19 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Lung Neoplasms
Keywords: Lung Cancer; HKI-272; Neratinib; Nerlynx
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — neratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Prior Tarceva or Iressa With EGFR Mutation (Experimental): HKI-272 administered to patients whose disease has progressed following > or = 12 weeks of treatment with Tarceva or Iressa and who have a tumor with an EGFR mutation demonstrated at screening
  Interventions: Drug: HKI-272
- Prior Tarceva or Iressa w/o EGFR Mutation (Experimental): HKI-272 administered to patients whose disease has progressed following > or = 12 weeks of treatment with Tarceva or Iressa and who have a tumor without an EGFR mutation demonstrated at screening
  Interventions: Drug: HKI-272
- No Prior EGFR Tyrosine Kinase Inhibitor Treatment (Experimental): HKI-272 administered to patients with no prior EGFR tyrosine kinase inhibitor treatment, adenocarcinoma, < or = 20 pack-year smoking history, and current non-smoker (no requirement for EGFR mutation)
  Interventions: Drug: HKI-272

INTERVENTIONS:
Drug: HKI-272 — 320mg or 240mg daily by mouth. The starting dose was reduced from 320mg to 240mg per amendment #1 to the protocol for subject safety and tolerability.
  Other Names: Neratinib

SUMMARY:
The purpose of this study is to learn whether HKI-272 is safe and effective in treating non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of NSCLC and current stage IIIB (with pleural effusion) or IV, not curable with conventional therapy. For Arm C, less than or equal to 20 pack-years smoking history and current non smoker. A pack year = number of packs of cigarettes smoked per day x years smoked.
* Progression following at least 12 weeks of treatment with Tarceva or Iressa. (Arms A and B only)
* ECOG (Eastern Cooperative Oncology Group) performance status of 0, 1, or 2 (not declining within past 2 weeks).
* Tumor sample available and adequate for analysis.
* At least one measurable target lesion.
* Adequate cardiac, kidney, and liver function
* Adequate blood counts

Exclusion Criteria:

* More than 3 prior cytotoxic chemotherapy treatments for relapsed or metastatic disease.
* Significant cardiac disease or dysfunction.
* Prior treatment with anthracyclines with cumulative dose of >400 mg/m^2.
* Active central nervous system metastases, as indicated by clinical symptoms and/or progressive growth.
* Use of Tarceva or Iressa within 14 days of treatment day 1 (Arms A and B only).
* Major surgery, chemotherapy, radiotherapy, investigational drugs, or other cancer therapy within 3 weeks of treatment day 1.
* Significant chronic or recent acute gastrointestinal disorder with diarrhea as a major symptom.
* Inability or unwillingness to swallow HKI-272 capsules.
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2005-12 (Actual); Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Puma, Study Director — Biotechnology
Locations (19):
- United States (11):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Midwestern Regional Medical Center, Zion, Illinois
  - Massachusetts General Hospital, Yawkey Center for Outpatient Care, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Memorial Sloan-Kettering, New York, New York
  - Carolinas Hematology-Oncology Associates, Charlotte, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Swedish Cancer Institute, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
- Institut Gustave Roussy, Villejuif, France
- Hungary (2):
  - Országos Korányi TBC és Pulmonológiai Intézet, Budapest
  - University of Debrecen, Debrecen
- Poland (4):
  - Akademia Medyczna W Gdansku, Gdansk
  - Mazowieckie Centrum Leczenia Chorób Płuc i Gruźlicy, Otwock
  - Wielkopolskie Centrum Chorób Płuc i Gruźlicy, Poznan
  - Dolnośląskie Centrum Chorób Płuc we Wrocławiu, Wroclaw
- Hospital Germans Trias I Puyol, Badalona, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Groups:
- Prior Tarceva or Iressa With EGFR Mutation: Patients whose disease has progressed following > or = 12 weeks of treatment with Tarceva or Iressa and who have a tumor with an EGFR mutation demonstrated at screening
  HKI-272: 320mg or 240mg daily by mouth. The starting dose was reduced from 320mg to 240mg per amendment #1 to the protocol for subject safety and tolerability.
- Prior Tarceva or Iressa w/o EGFR Mutation: Patients whose disease has progressed following > or = 12 weeks of treatment with Tarceva or Iressa and who have a tumor without an EGFR mutation demonstrated at screening
  HKI-272: 320mg or 240mg daily by mouth. The starting dose was reduced from 320mg to 240mg per amendment #1 to the protocol for subject safety and tolerability.
- No Prior EGFR Tyrosine Kinase Inhibitor Treatment: Patients with no prior EGFR tyrosine kinase inhibitor treatment, adenocarcinoma, < or = 20 pack-year smoking history, and current non-smoker (no requirement for EGFR mutation)
  HKI-272: 320mg or 240mg daily by mouth. The starting dose was reduced from 320mg to 240mg per amendment #1 to the protocol for subject safety and tolerability.
Period: Overall Study
Arm/Group | Prior Tarceva or Iressa With EGFR Mutation | Prior Tarceva or Iressa w/o EGFR Mutation | No Prior EGFR Tyrosine Kinase Inhibitor Treatment
Started | 91 | 48 | 28
Completed | 0 | 0 | 0
Not Completed | 91 | 48 | 28
Not completed — Death | 1 | 1 | 1
Not completed — Adverse Event | 6 | 4 | 1
Not completed — Physician Decision | 2 | 1 | 1
Not completed — Withdrawal by Subject | 3 | 1 | 1
Not completed — Disease Progression | 72 | 37 | 23
Not completed — Symptomatic Deterioration | 6 | 3 | 1
Not completed — Hospitalization | 1 | 0 | 0
Not completed — Concomitant Radiotherapy | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prior Tarceva or Iressa With EGFR Mutation | Prior Tarceva or Iressa w/o EGFR Mutation | No Prior EGFR Tyrosine Kinase Inhibitor Treatment | Total
Number analyzed (Participants) | 91 | 48 | 28 | 167
Age, Customized [Count of Participants; unit: Participants]
  < 60 years | 45 | 24 | 13 | 82
  >= 60 years | 46 | 24 | 15 | 85
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 26 | 18 | 118
  Male | 17 | 22 | 10 | 49

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate for Neratinib in Patients With Non-small Cell Lung Cancer
Description: Objective response rate as reported by Independent Assessment (radiographic review by independent radiologists) per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.0: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; and Non-PD for non-target lesions, and no new lesions.
Time Frame: From first dose date to progression/death or last tumor assessment, up to three years.
Population: modified ITT: Subjects who were randomized and who had taken at least 1 dose of neratinib; equivalent to the safety population
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Prior Tarceva or Iressa With EGFR Mutation | Prior Tarceva or Iressa w/o EGFR Mutation | No Prior EGFR Tyrosine Kinase Inhibitor Treatment
Number analyzed (Participants) | 91 | 48 | 28
percentage of participants | 3.3 [0.9 to 8.3] | 0 [0 to 6.05] | 3.6 [0.18 to 15.85]

2. Secondary Outcome: Clinical Benefit Rate for Neratinib in Patients With Non-small Cell Lung Cancer
Description: Clinical benefit rate is the percentage of patients with Partial or Complete Response, or with Stable Disease >= 12 Weeks per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.0: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; and Non-PD for non-target lesions, and no new lesions; Stable Disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: From first dose date to progression/death or last tumor assessment, up to three years.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Prior Tarceva or Iressa With EGFR Mutation | Prior Tarceva or Iressa w/o EGFR Mutation | No Prior EGFR Tyrosine Kinase Inhibitor Treatment
Number analyzed (Participants) | 91 | 48 | 28
percentage of participants | 9.9 [5.26 to 16.62] | 6.3 [1.73 to 15.37] | 10.7 [2.98 to 25.42]

3. Secondary Outcome: Duration of Response for Neratinib in Patients With Non-small Cell Lung Cancer
Description: Measured from the time at which measurement criteria were first met for CR or PR (whichever status was recorded first), until the date of first recurrence, PD, or death was objectively documented, taking as a reference for PD the smallest measurements recorded since enrollment, per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.0: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; and Non-PD for non-target lesions, and no new lesions.
Time Frame: From start date of response to first PD, assessed up to three years after the first randomization.
Population: Number of subjects with PR or higher response.
Measure: Median (90% Confidence Interval); unit: weeks
Arm/Group | Prior Tarceva or Iressa With EGFR Mutation | Prior Tarceva or Iressa w/o EGFR Mutation | No Prior EGFR Tyrosine Kinase Inhibitor Treatment
Number analyzed (Participants) | 3 | 0 | 1
weeks | 54.1 [17.9 to 54.1] |  | 28.7 [NA to NA] — Insufficient number of participants with events.

4. Secondary Outcome: Progression Free Survival for Neratinib in Patients With Non-small Cell Lung Cancer
Description: Defined as the interval from the date of randomization until the first date on which recurrence or progression, or death due to any cause, is documented, censored at the last assessable evaluation or at the initiation of new anticancer therapy. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v 1.0 as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From first dose date to progression/death, assessed up to three years.
Measure: Median (90% Confidence Interval); unit: weeks
Arm/Group | Prior Tarceva or Iressa With EGFR Mutation | Prior Tarceva or Iressa w/o EGFR Mutation | No Prior EGFR Tyrosine Kinase Inhibitor Treatment
Number analyzed (Participants) | 91 | 48 | 28
weeks | 15.3 [11.9 to 15.7] | 16.1 [15.0 to 23.9] | 9.3 [6.4 to 18.9]

ADVERSE EVENTS:
Time Frame: First dose through 28 days after last dose, assessed up to three years.
Arm/Group | Prior Tarceva or Iressa With EGFR Mutation | Prior Tarceva or Iressa w/o EGFR Mutation | No Prior EGFR Tyrosine Kinase Inhibitor Treatment
Serious Adverse Events (participants affected / at risk) | 33/91 | 21/48 | 14/28
Other Adverse Events (participants affected / at risk) | 91/91 | 46/48 | 26/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prior Tarceva or Iressa With EGFR Mutation (N=91) | Prior Tarceva or Iressa w/o EGFR Mutation (N=48) | No Prior EGFR Tyrosine Kinase Inhibitor Treatment (N=28)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Acute abdomen (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 2
Nausea (Gastrointestinal disorders) | 4 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 2
Fatigue (General disorders) | 0 | 0 | 1
General physical health deterioration (General disorders) | 5 | 3 | 3
Hyperthermia (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1
Unevaluable event (General disorders) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 3 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0
Cerebral venous thrombosis (Nervous system disorders) | 1 | 0 | 0
Coma (Nervous system disorders) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0
Radicular syndrome (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Speech disorder (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prior Tarceva or Iressa With EGFR Mutation (N=91) | Prior Tarceva or Iressa w/o EGFR Mutation (N=48) | No Prior EGFR Tyrosine Kinase Inhibitor Treatment (N=28)
Anaemia (Blood and lymphatic system disorders) | 11 | 9 | 8
Lymphopenia (Blood and lymphatic system disorders) | 11 | 4 | 8
Abdominal distension (Gastrointestinal disorders) | 6 | 2 | 4
Abdominal pain (Gastrointestinal disorders) | 36 | 14 | 5
Abdominal pain upper (Gastrointestinal disorders) | 8 | 2 | 1
Constipation (Gastrointestinal disorders) | 10 | 4 | 4
Diarrhoea (Gastrointestinal disorders) | 85 | 41 | 25
Dry mouth (Gastrointestinal disorders) | 1 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 2 | 3
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 2
Flatulence (Gastrointestinal disorders) | 5 | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 3 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 52 | 24 | 16
Vomiting (Gastrointestinal disorders) | 36 | 14 | 9
Asthenia (General disorders) | 22 | 9 | 6
Chest pain (General disorders) | 12 | 7 | 2
Fatigue (General disorders) | 36 | 19 | 7
Oedema peripheral (General disorders) | 2 | 3 | 1
Pyrexia (General disorders) | 11 | 6 | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 3
Folliculitis (Infections and infestations) | 1 | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 1 | 4
Pulpitis dental (Infections and infestations) | 0 | 0 | 2
Rhinitis (Infections and infestations) | 2 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 6 | 1
Alanine aminotransferase increased (Investigations) | 7 | 1 | 3
Amylase increased (Investigations) | 6 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 4 | 2 | 3
Blood alkaline phosphatase increased (Investigations) | 3 | 4 | 4
Blood creatinine increased (Investigations) | 3 | 2 | 2
Blood lactate dehydrogenase increased (Investigations) | 2 | 4 | 4
Gamma-glutamyltransferase increased (Investigations) | 5 | 5 | 2
Protein total decreased (Investigations) | 0 | 3 | 2
Weight decreased (Investigations) | 7 | 8 | 4
Cell death (Metabolism and nutrition disorders) | 4 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 35 | 16 | 11
Dehydration (Metabolism and nutrition disorders) | 15 | 6 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 3 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 4 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 3 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 6 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 7 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 4 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 1 | 1
Dizziness (Nervous system disorders) | 11 | 4 | 0
Dysgeusia (Nervous system disorders) | 4 | 2 | 4
Headache (Nervous system disorders) | 15 | 8 | 4
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 2
Neuralgia (Nervous system disorders) | 0 | 0 | 3
Paraesthesia (Nervous system disorders) | 0 | 2 | 2
Confusional state (Psychiatric disorders) | 2 | 3 | 0
Depression (Psychiatric disorders) | 6 | 3 | 2
Disorientation (Psychiatric disorders) | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 6 | 2 | 2
Haematuria (Renal and urinary disorders) | 3 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 5 | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 | 13 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 | 2 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 15 | 7 | 5
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 8 | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 16 | 8 | 9
Skin fissures (Skin and subcutaneous tissue disorders) | 2 | 2 | 2
Thrombosis (Vascular disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less